CLINICAL TRIAL: NCT00503139
Title: Enbrel Special Use Result Surveillance
Brief Title: Study Evaluating the Safety and Efficacy of Enbrel (Etanercept) in Japan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-4426; B1801045 (Other: Alias Study Number)
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Enbrel (etanercept) — Enbrel 10 to 25 mg twice a week subcutaneous injection

SUMMARY:
The special use-results surveillance is conducted in patients who have never been treated with Enbrel and in whom its long-term therapy may be instituted in the actual setting of use after marketing with the following objectives: 1. To examine the safety of long-term use of Enbrel including the occurrence of malignant tumors. 2. To confirm the efficacy of Enbrel in the long-term use.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Patients with rheumatoid arthritis (RA) who fulfill all of the following

1. Patients who are refractory to the treatment.
2. Patients who have never been treated with Enbrel and in whom its long-term therapy may be instituted.
3. Patients without a history of or concurrent malignant tumors.

Exclusion Criteria:

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital and Rheumatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2007-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Hokkaido University Hospital, Sapporo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-4426&StudyName=Study%20Evaluating%20the%20Safety%20and%20Efficacy%20of%20Enbrel%20%28Etanercept%29%20in%20Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept (Genetical Recombination): Participants who received etanercept (genetical recombination) 10 to 25 mg once daily (twice weekly) or 25 to 50 mg once daily (once weekly) subcutaneously.
Period: Overall Study
Arm/Group | Etanercept (Genetical Recombination)
Started | 684
Completed | 676
Not Completed | 8
Not completed — Case Report Forms were not collected | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 676
Age, Customized [Number; unit: Participants]
  <65 years | 454
  >=65 years | 222
Gender [Count of Participants; unit: Participants]
  Female | 559
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Safety Analysis Population of Etanercept
Time Frame: 3 years
Population: The safety analysis population (N = number of participants evaluated) consisted of the participants who received etanercept for rheumatoid arthritis because of an inadequate response to the conventional therapies and had no history of or concurrent malignant tumors.
Measure: Number; unit: Participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 676
Participants
  Within 6 months | 676
  6 to 12 months | 561
  Within 1 year | 676
  1 to 2 years | 475
  2 to 3 years | 372
  3 years or more | 176

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Etanercept
Description: Adverse events are all unfavorable events, including clinically problematic abnormal changes in laboratory test values, which develop in participants after the administration of Etanercept, irrespective of causal relationship to Etanercept. The causal relationship between an adverse event and Etanercept was evaluated by the sponsor.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 676
Participants
  Within 6 months (N=676) | 117
  6 to 12 months (N=561) | 84
  Within 1 year (N=676) | 184
  1 to 2 years (N=475) | 90
  2 to 3 years (N=372) | 43
  3 years or more (N=176) | 1

3. Primary Outcome: Number of Participants With Serious Treatment Related Adverse Events of Etanercept
Description: Serious treatment-related adverse events are defined as any events that lead to death, life-threatening, hospitalization or prolonged hospitalization, a permanent or remarkable disorder/dysfunction, congenital anomaly/congenital deficiency, or other medically significant events or disorder.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 676
Participants
  Within 6 months (N = 676) | 12
  6 to 12 months (N = 561) | 17
  Within 1 year (N = 676) | 29
  1 to 2 years (N = 475) | 24
  2 to 3 years (N = 372) | 13
  3 years or more (N = 176) | 0

4. Primary Outcome: Number of Participants With Unlisted Treatment Related Adverse Events of Etanercept
Description: Adverse events are all unfavorable events, including clinically problematic abnormal changes in laboratory test values, which develop in participants after the administration of Etanercept, irrespective of causal relationship to Etanercept. The causal relationship between an adverse event and Etanercept was evaluated by the sponsor. Unlisted treatment related adverse events were confirmed with listed adverse drug reactions specified in Japanese package insert.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 676
Participants | 16

5. Primary Outcome: European League Against Rheumatism (EULAR) Disease Activity Score (DAS) 28 Improvement (4/Erythrocyte Sedimentation Rate: ESR)
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment). Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission.
Time Frame: 2 years
Population: The efficacy analysis population (N = number of participants evaluated) consisted of the participants in whom DAS28 (4/ESR) was calculated. The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 583
percentage of participants
  At 6 months (N = 533) | 84.05 [80.66 to 87.06]
  At 1 year (N = 566) | 82.51 [79.12 to 85.55]
  At 1.5 years (N = 576) | 79.69 [76.17 to 82.90]
  At 2 years (N = 577) | 81.98 [78.59 to 85.03]

6. Secondary Outcome: Modified Health Assessment Questionnaire (mHAQ) Score
Description: Modified Health Assessment Questionnaire-(mHAQ): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: 2 years
Population: The efficacy analysis population (N = number of participants evaluated) consisted of the participants in whom mHAQ was calculated. The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 583
Score
  At Baseline (N = 583) | 0.82 (0.64)
  At 6 months (N = 490) | 0.45 (0.58)
  At 1 year (N = 520) | 0.46 (0.61)
  At 1.5 years (N = 526) | 0.45 (0.61)
  At 2 years (N = 531) | 0.46 (0.60)
Statistical Analysis 1: Comparison: Etanercept (Genetical Recombination); The null hypothesis was that mHAQ scores at 6 months, 1 year, 1.5 years, and 2 years were equal to the baseline score; Test type: Superiority or Other; p < 0.001, t-test, 1 sample; A two-sided t-test was performed to test the hypothesis

7. Secondary Outcome: Visual Analog Fatigue Scale (VAFS)
Description: Participants assessed their fatigue using a 0 - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: 2 years
Population: The efficacy analysis population (N = number of participants evaluated) consisted of the participants in whom VAS Fatigue was calculated. The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 583
Score
  At Baseline (N = 583) | 49.1 (27.1)
  At 6 months (N = 477) | 26.1 (22.6)
  At 1 year (N = 509) | 25.2 (22.8)
  At 1.5 years (N = 513) | 25.3 (23.2)
  At 2 years (N = 518) | 26.0 (23.8)
Statistical Analysis 1: Comparison: Etanercept (Genetical Recombination); The null hypothesis was that VAS Fatigue scores at 6 months, 1 year, 1.5 years, and 2 years were equal to the baseline score; Test type: Superiority or Other; p < 0.001, t-test, 1 sample; A two-sided t-test was performed to test the hypothesis

8. Secondary Outcome: European League Against Rheumatism (EULAR) Disease Activity Score (DAS) 28 Improvement (3/Erythrocyte Sedimentation Rate: ESR)
Description: DAS28-3 (ESR) was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count and ESR (mm/hour). Total score range: 0-9.4, higher score=more disease activity. DAS28-3 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (ESR) <2.6 = remission.
Time Frame: 2 years
Population: The efficacy analysis population (N = number of participants evaluated) consisted of the participants in whom DAS28 (3/ESR) was calculated. The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept (Genetical Recombination)
Number analyzed (Participants) | 583
percentage of participants
  At 6 months (N = 533) | 81.80 [78.26 to 84.99]
  1 year (N = 566) | 81.10 [77.62 to 84.24]
  1.5 years (N = 576) | 79.69 [76.17 to 82.90]
  2 years (N = 577) | 80.42 [76.94 to 83.58]

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study
Arm/Group | Etanercept (Genetical Recombination)
Serious Adverse Events (participants affected / at risk) | 77/676
Other Adverse Events (participants affected / at risk) | 261/676
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (Genetical Recombination) (N=676)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 2 (2)
Skin bacterial infection (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bone tuberculosis (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Atypical mycobacterial infection (Infections and infestations) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Senile dementia (Nervous system disorders) | 1 (1)
Vertebral artery occlusion (Nervous system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
Aortic dissection rupture (Vascular disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Granulocyte count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Renal stone removal (Surgical and medical procedures) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (Genetical Recombination) (N=676)
Acute sinusitis (Infections and infestations) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 19 (23)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 4 (4)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4)
Hepatitis C (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 11 (11)
Influenza (Infections and infestations) | 2 (2)
Nail candida (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 25 (27)
Onychomycosis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (3)
Otitis media (Infections and infestations) | 2 (2)
Parotitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 7 (10)
Pneumonia (Infections and infestations) | 6 (6)
Pyelonephritis (Infections and infestations) | 2 (2)
Rash pustular (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (7)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 4 (5)
Convulsion (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (5)
Sciatica (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1)
Erythema of eyelid (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 19 (24)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 7 (7)
Submaxillary gland enlargement (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 25 (30)
Hepatic steatosis (Hepatobiliary disorders) | 3 (4)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 5 (5)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 9 (11)
Erythema (Skin and subcutaneous tissue disorders) | 8 (10)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 13 (15)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Skin chapped (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (7)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Injection site pain (General disorders) | 4 (4)
Injection site reaction (General disorders) | 30 (31)
Malaise (General disorders) | 4 (4)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 9 (11)
Foreign body reaction (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (3)
Blood urea increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 4 (4)
Laboratory test abnormal (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 7 (7)
Platelet count decreased (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 7 (7)
Blood beta-D-glucan increased (Investigations) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Antinuclear antibody positive (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 6 (6)
DNA antibody positive (Investigations) | 1 (1)
Cell marker increased (Investigations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.